CLINICAL TRIAL: NCT00064987
Title: Role of FSH in Human Gonadal Development
Brief Title: Follicle Stimulating Hormone (FSH) to Improve Testicular Development in Men With Hypogonadism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was at a standstill. We are currently preparing our results for publication.
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, William Crowley, Principle Investigator, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U54HD028138-457; U54HD028138 (NIH)
Record Dates: First submitted 2003-07-16; First posted 2003-07-17 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Hypogonadism; Kallmann Syndrome
Keywords: Male reproduction hormones; Hypogonadotropic hypogonadism; FSH; LH; GnRH
MeSH Terms: conditions — Hypogonadism; Kallmann Syndrome | interventions — Gonadotropin-Releasing Hormone; Follicle Stimulating Hormone; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (FSH) (Experimental): Patients in Group 1 will receive subcutaneous follicle stimulating hormone (FSH) injections daily, titrated to achieve a FSH level of 4-8 IU/L, for 4 months. Patients will then receive gonadotropin releasing hormone (GnRH) therapy for 18 months. GnRH will be administered via a portable infusion pump at 2-hour intervals to stimulate endogenous LH secretion.
  Interventions: Procedure: Testicular biopsy; Drug: gonadotropin releasing hormone (GnRH); Drug: follicle stimulating hormone (FSH)
- Group 2 (GnRH) (Active Comparator): Patients in Group 2 will receive gonadotropin releasing hormone (GnRH) therapy for 18 months. GnRH will be administered via a portable infusion pump at 2-hour intervals to stimulate endogenous LH secretion. Patients in Group 2 will not receive prior FSH administration.
  Interventions: Procedure: Testicular biopsy; Drug: gonadotropin releasing hormone (GnRH)

INTERVENTIONS:
Procedure: Testicular biopsy — Outpatient surgical procedure.
Drug: gonadotropin releasing hormone (GnRH) — Pulsatile GnRH (25 ng/kg per bolus every two hours via microinfusion pump titrated to reach normal serum testosterone levels)
Drug: follicle stimulating hormone (FSH) — 75 IU subcutaneous injection daily for four months.
  Other Names: Gonal-F
  Arms: Group 1 (FSH)

SUMMARY:
Men with idiopathic hypogonadotropic hypogonadism (IHH, Kallmann Syndrome) may have small testicular size, low testosterone levels, no history of puberty, and infertility. These men lack a hormone called gonadotropin releasing hormone (GnRH) that stimulates the development and maturation of the testes. This study will investigate the impact of hormonal treatments on men with IHH. The goal of hormonal therapy is to maximize the potential fertility in these individuals.

DETAILED DESCRIPTION:
Though steroid output of the testes is minimal during childhood, important changes take place that impact spermatogenic potential. Specifically, the number of Sertoli cells increases until testosterone secretion rises during puberty. In animal models, the proliferation of Sertoli cells appears to be regulated by follicle stimulating hormone (FSH) even though FSH levels in childhood are relatively low. At puberty, the number of Sertoli cells becomes fixed; however, the existing cell population then undergoes functional maturation. This switch from proliferation to maturation of Sertoli cells appears to result from rising levels of intratesticular testosterone.

FSH deficiency during testicular development results in decreased numbers of Sertoli cells, even if physiologic hormonal replacement therapy is introduced in adolescence or adulthood. The number of mature Sertoli cells appears to correlate with testicular size, sperm count, and future fertility. An improved understanding of the specific roles of FSH, luteinizing hormone (LH), and testosterone in testicular development may have direct clinical applications in the treatment of male infertility. This study will define the role of FSH in stimulating Sertoli cell proliferation in the human male.

Patients in this study will be randomized to receive either FSH and GnRH (Group 1) or GnRH alone (Group 2). Patients in Group 1 will receive subcutaneous FSH injections daily, titrated to achieve a FSH level of 4-8 IU/L, for 4 months. Patients will then receive GnRH therapy for 18 months. GnRH will be administered via a portable infusion pump at 2-hour intervals to stimulate endogenous LH secretion. Patients in Group 2 will receive the same regimen of exogenous GnRH for 18 months without prior FSH administration.

All patients will undergo an initial assessment that includes an overnight 12-hour frequent blood sampling study, testicular ultrasound, and testicular biopsy. Patients will be followed through monthly study visits with blood tests and seminal fluid analysis. Patients will also have serial testicular ultrasounds to measure testicular growth. Patients in Group 1 will also have a second frequent blood sampling to measure LH, FSH, and testosterone and to confirm the absence of LH pulses.

ELIGIBILITY:
Inclusion Criteria

* no history of spontaneous puberty
* clinical hypogonadism
* infantile testes (< 3 ml)
* no reproductive hormone therapy except testosterone
* Complete absence of normal LH pulses during 12-hour baseline frequent blood sampling and serum testosterone < 100 ng/dl
* Normal testing of the anterior pituitary gland
* Negative MRI of the hypothalamic-pituitary area

Exclusion Criteria

* Prior therapy with gonadotropins (FSH, hCG, or GnRH)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William F Crowley, Jr., MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Pitteloud N, Hayes FJ, Dwyer A, Boepple PA, Lee H, Crowley WF Jr. Predictors of outcome of long-term GnRH therapy in men with idiopathic hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 2002 Sep;87(9):4128-36. doi: 10.1210/jc.2002-020518. PMID 12213860
- [Background] Pitteloud N, Hayes FJ, Boepple PA, DeCruz S, Seminara SB, MacLaughlin DT, Crowley WF Jr. The role of prior pubertal development, biochemical markers of testicular maturation, and genetics in elucidating the phenotypic heterogeneity of idiopathic hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 2002 Jan;87(1):152-60. doi: 10.1210/jcem.87.1.8131. PMID 11788640
- [Background] Hayes FJ, Pitteloud N, DeCruz S, Crowley WF Jr, Boepple PA. Importance of inhibin B in the regulation of FSH secretion in the human male. J Clin Endocrinol Metab. 2001 Nov;86(11):5541-6. doi: 10.1210/jcem.86.11.8031. PMID 11701733
- [Background] Kumar PA, Pitteloud N, Andrews PA, Dwyer A, Hayes F, Crowley WF Jr, Dym M. Testis morphology in patients with idiopathic hypogonadotropic hypogonadism. Hum Reprod. 2006 Apr;21(4):1033-40. doi: 10.1093/humrep/dei444. Epub 2006 Jan 5. PMID 16396935
- [Derived] Dwyer AA, Sykiotis GP, Hayes FJ, Boepple PA, Lee H, Loughlin KR, Dym M, Sluss PM, Crowley WF Jr, Pitteloud N. Trial of recombinant follicle-stimulating hormone pretreatment for GnRH-induced fertility in patients with congenital hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 2013 Nov;98(11):E1790-5. doi: 10.1210/jc.2013-2518. Epub 2013 Sep 13. PMID 24037890

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were deemed ineligible for the study. One subject was lost to follow up before being assigned to Group 1 or Group 2.
Groups:
- Group 1 (FSH): Patients in Group 1 will receive subcutaneous FSH injections daily, titrated to achieve a FSH level of 4-8 IU/L, for 4 months. Patients will then receive GnRH therapy for 18 months. GnRH will be administered via a portable infusion pump at 2-hour intervals to stimulate endogenous LH secretion.
- Group 2 (GnRH): Patients in Group 2 will receive GnRH therapy for 18 months. GnRH will be administered via a portable infusion pump at 2-hour intervals to stimulate endogenous LH secretion. Patients in Group 2 will not receive prior FSH administration.
Period: Overall Study
Arm/Group | Group 1 (FSH) | Group 2 (GnRH)
Started | 10 | 6
Completed | 7 | 6
Not Completed | 3 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (FSH) | Group 2 (GnRH) | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: LH
Description: Average Luteinizing Hormone levels after treatment.
Time Frame: month 4 of GnRH treatment
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Group 1 (FSH) | Group 2 (GnRH)
Number analyzed (Participants) | 7 | 6
IU/L | 12.7 (.5) | 16.5 (.7)

2. Primary Outcome: FSH
Description: Average Follicle Stimulating Hormone levels after treatment.
Time Frame: month 4 of GnRH treatment
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Group 1 (FSH) | Group 2 (GnRH)
Number analyzed (Participants) | 7 | 6
IU/L | 9.9 (.4) | 15.6 (1.1)

3. Primary Outcome: Testosterone
Description: Average Testosterone levels after treatment.
Time Frame: month 4 of GnRH treatment
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Group 1 (FSH) | Group 2 (GnRH)
Number analyzed (Participants) | 7 | 6
ng/dL | 299 (14) | 330 (15)

4. Primary Outcome: Inhibin B
Description: Average Inhibin B Levels after treatment.
Time Frame: month 4 of GnRH treatment
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Group 1 (FSH) | Group 2 (GnRH)
Number analyzed (Participants) | 7 | 6
pg/mL | 110 (5) | 74 (4)

5. Primary Outcome: Testicular Size (Volume)
Description: Average testicular volume after treatment.
Time Frame: at baseline and month 4 of GnRH treatment
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Group 1 (FSH) | Group 2 (GnRH)
Number analyzed (Participants) | 7 | 6
mL
  Before Treatment | 1.1 (.2) | .8 (.2)
  After Treatment | 9.3 (1.7) | 6.6 (1.3)

6. Primary Outcome: Sperm Count
Description: Average sperm count after treatment.
Time Frame: month 4 of GnRH treatment
Measure: Mean (Standard Deviation); unit: 10^6 sperms/mL
Arm/Group | Group 1 (FSH) | Group 2 (GnRH)
Number analyzed (Participants) | 7 | 6
10^6 sperms/mL | 5.8 (2.3) | 2.6 (1.5)

7. Secondary Outcome: Fertility
Description: Participants actively seeking to conceive.
Time Frame: 24 months
Population: Four subjects in Group 1 and two subjects in Group 2 were actively trying to conceive. Fertility was not tracked in subjects not trying to conceive.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (FSH) | Group 2 (GnRH)
Number analyzed (Participants) | 4 | 2
Participants | 4 | 1

ADVERSE EVENTS:
Arm/Group | Group 1 (FSH) | Group 2 (GnRH)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No